CLINICAL TRIAL: NCT03425006
Title: Phase II Study of Pembrolizumab and Itacitinib (INCB039110) for First Line Treatment of Metastatic Non-Small Cell Lung Cancer Expressing PD-L1
Brief Title: Pembrolizumab and Itacitinib (INCB039110) for Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC# 09517; IRB# 828910
Record Dates: First submitted 2018-01-22; First posted 2018-02-07 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — itacitinib; INCB039110; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Itacitinib and Pembrolizumab (Experimental)
  Interventions: Drug: Itacitinib; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Itacitinib — a JAK 1 selective small molecule inhibitor
  Other Names: INCB039110
Biological: Pembrolizumab — a highly selective humanized monoclonal antibody (mAb)

SUMMARY:
This is a single center, single arm phase 2 study to establish the safety and efficacy of itacitinib (also known as INCB039110) administered in combination with pembrolizumab in patients with metastatic PD-L1 positive non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* 1. Stage IV or metastatic non-small cell lung cancer (NSCLC)
* 2. Provide written informed consent for the trial.
* 3. Patients ≥ 18 years of age
* 4. Tumor PD-L1≥ 50% as assessed by the PD-L1 IHC 22C3 pharmDx assay (Dako North America).
* 5. Subject must have adequate tumor burden at a safely accessible site for biopsy. NOTE: If sites chosen for biopsy were previously irradiated, there must be evidence of tumor growth/viable tumor as assessed by the investigator.
* 6. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* 7. ECOG performance status 0 or 1
* 8. Adequate Organ Function Laboratory Values: Absolute neutrophil count (ANC) ≥1,250/mcL; Platelets ≥100,000/mcL; Hemoglobin ≥9 g/dL or ≥5.6 mmol/L; Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥50 mL/min for subject with creatinine levels > 1.5 X institutional ULN; Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN; AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* 9. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

* 1. Sensitizing mutations in Epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) or ROS1 proto-oncogene receptor tyrosine kinase (ROS1) translocations
* 2. Currently participating in or has participated in a study of an investigational agent or anticipated use of an investigational device within 4 weeks of the first dose of study treatment.
* 3. Untreated symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis.
* 4. Received prior systemic cytotoxic chemotherapy, biologic therapy, targeted therapy or immunotherapy for incurable (metastatic) NSCLC.
* 5. Diagnosis of immunodeficiencywithin 7 days prior to eligibility confirmation by the physician-investigator.
* 6. Prior monoclonal antibodies used for the treatment of NSCLC within 4 weeks prior to eligibility confirmation by the physician-investigator, or individuals who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* 7. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, non-invasive bladder tumors, or in situ cervical cancer
* 8. 8. Active autoimmune disease requiring systemic immunosuppressive treatment within the past 3 months prior to eligibility confirmation by the physician-investigator. Subjects that require intermittent use of steroid-containing bronchodilators or local steroid injections or topical steroid medications are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome are not excluded from the study.
* 9. Interstitial lung disease or history of pneumonitis that has required oral or IV steroids
* 10. Active infection requiring systemic therapy with IV antibiotics
* 11. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* 12. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* 13. Pregnant or breastfeeding women
* 14. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4).
* 15. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* 16. Known active Hepatitis B (e.g., HBsAg positive or HBV DNA detectable) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* 17. Anticipated receipt of any live vaccine within 30 days prior to the first dose of trial treatment.

Note: For the purposes of determining eligibility above, enrollment is defined as the date of subject consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Langer, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Itacitinib and Pembrolizumab: Dose and Route of Administration
  * Itacitinib: 200mg PO (extended release formulation)
  * Pembrolizumab: 200mg IV infusion over 30 minutes Regimen
  * Treatment = 3 week (Q3W) dosing cycles
  * Itacitinib: Once daily for Cycle 3 and Cycle 4 (up to 6 weeks)
  * Pembrolizumab: Q3 week cycles of treatment beginning at Day 1
Period: Overall Study
Arm/Group | Itacitinib and Pembrolizumab
Started | 23
Completed | 20
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Itacitinib and Pembrolizumab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Response at 12 Weeks According to RECIST 1.1 for the Combination of Pembrolizumab and Itacitinib Among Patients With Previously Untreated, PD-L1 Positive Metastatic NSCLC.
Description: Responses will be compared subject's baseline assessment and historical controls using pembrolizumab monotherapy.
Time Frame: 12 weeks
Population: Of the 23 subjects enrolled, 2 subjects were not included in analysis because they did not receive Itacitinib due to pembrolizumab toxicity or subject withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib and Pembrolizumab
Number analyzed (Participants) | 21
Participants | 13

2. Primary Outcome: Number of Subjects With Toxicities (CTCAE v5.0 Scoring) of Pembrolizumab and Itacitinib in Patients With Previously Untreated, PD-L1 Positive Metastatic NSCLC
Description: Number of subjects treated with the combination.
Time Frame: 16 weeks
Population: Of the 23 subjects enrolled, 3 subjects were not included in analysis because they only received pembrolizumab and not itacitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib and Pembrolizumab
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: Number of Participants Who Had a Progression Free Survival (PFS) Treated With Pembrolizumab and Itacitinib.
Description: Number of participants who remained progression free at week 12
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib and Pembrolizumab
Number analyzed (Participants) | 23
Participants | 20

4. Secondary Outcome: Number of Participants Treated With Pembrolizumab and Itacitinib, Who Had a Minimum Duration of Response (DOR) of 12 Weeks.
Time Frame: 12 weeks
Population: Of the 23 subjects enrolled, 2 subjects were not included in analysis because they did not receive Itacitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib and Pembrolizumab
Number analyzed (Participants) | 21
Participants | 13

5. Secondary Outcome: Overall Survival (OS) for Subjects Treated With Pembrolizumab and Itacitinib.
Description: Number of subjects treated with pembrolizumab and itacitinib that survived to week 16.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib and Pembrolizumab
Number analyzed (Participants) | 23
Participants | 23

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Itacitinib and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itacitinib and Pembrolizumab (N=23)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Hemorrhagic brain metastasis
Seizure (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Vasogenic edema
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itacitinib and Pembrolizumab (N=23)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 7 (9)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 8 (8)
Fever (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 3 (3)
Weight gain (Investigations) | 4 (4)
Weight loss (Investigations) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (6)
Insomnia (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT03425006/Prot_SAP_000.pdf